CLINICAL TRIAL: NCT06384196
Title: Identity-Based Transdiagnostic Therapy for Young People With Anxiety and Depression: Engagement, Efficacy, and Predictors of Outcome
Brief Title: Identity-Based Transdiagnostic Therapy for Young People With Anxiety and Depression
Acronym: IBTTYOUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Badalona Serveis Assistencials (Other); Nou Barris Mental Health Center (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Full Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2022-138902OB-I00
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety
Keywords: Young Adult; Virtual Reality; Self-identity; Sense of identity; Psychological Conflict; Self-concept; Self-assessment; Metacognitive Awareness; Cognitive Reflection; Personal Satisfaction; Patient Satisfaction; Psychological Well-Being; Therapeutic Alliance; Treatment Outcome
MeSH Terms: conditions — Depression; Anxiety Disorders; Personal Satisfaction; Patient Satisfaction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The main study of this project proposal is a multi-center, single-blind, parallel-group randomized clinical trial (RCT) conducted in Catalonia (Spain).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Identity-Based Transdiagnostic Therapy (IBTT) (Experimental): IBTT is based on Personal Construct Therapy enhanced with Virtual Reality. In this version, psychotherapy focuses on identity conflicts and processes using an immersive exploration of self and others. After some observational evidence, this is the first study to test the efficacy of this innovative approach rigorously.
  Interventions: Behavioral: Identity-Based Transdiagnostic Therapy (IBTT)
- Unified Protocol (UP) (Active Comparator): The UP is a transdiagnostic psychotherapy for anxiety and/or depression based on Cognitive-Behavioral Therapy (CBT). Several previous studies provide substantive evidence for the efficacy of the UP for these disorders.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Identity-Based Transdiagnostic Therapy (IBTT) — In this study, IBTT is applied in 16, one-hour weekly sessions based on contemporary constructivist psychotherapy enhanced with the technological platform EYME-Explore Your Meanings to enable the immersive exploration of the patient's self-identity. Although it could be applied to other populations, IBTT has been designed to improve the mental health of late adolescents and young people.
  Arms: Identity-Based Transdiagnostic Therapy (IBTT)
Behavioral: Unified Protocol — In this study, the UP is applied in 16, one-hour weekly sessions based on contemporary cognitive and behavioral techniques.
  Arms: Unified Protocol (UP)

SUMMARY:
Depression and anxiety are the most prevalent mental disorders among both the general population and young adults, and transdiagnostic treatments for these patients are mostly based on cognitive-behavioral therapy (CBT). Based on common (transdiagnostic) principles of treatment (e.g., emotional exposure), these approaches have proliferated and demonstrated their efficacy in comparison to disorder-specific treatments. Although there are a few transdiagnostic approaches for children and adolescents, it was not possible to not find anyone targeting young people. For this reason, the investigators proposed the Identity-Based Transdiagnostic Therapy (IBTT) as a new treatment modality ideally created to address the challenge of improving the outcomes of psychotherapy for young adults with anxiety and/or depression. The IBTT is a psychological treatment for emotional disorders specifically designed for the youths in terms of their attitudes to treatment (attractiveness, engagement), and highly personalized to their construal of self and others. This project will allow testing the hypothesis that a novel brief psychotherapeutic intervention, IBTT, will be more efficacious in the treatment of the anxiety and/or depression of young adults than the well-established CBT-based Unified Protocol.

DETAILED DESCRIPTION:
Depression and anxiety are the most prevalent mental disorders among both the general population and young adults, and transdiagnostic treatments for these patients are mostly based on cognitive-behavioral therapy (CBT). One reason for their emergence is the observation of common psychological processes (e.g., negative affectivity) among emotional disorders that outweigh differences between specific disorders. Relatedly, in favor of a transdiagnostic approach, there is the more pragmatic argument of the high comorbidity among these disorders, making the consecutive application of specific manuals a barrier to evidence-based practice in the real world. Based on common (transdiagnostic) principles of treatment (e.g., emotional exposure), these approaches have proliferated and demonstrated their efficacy in comparison to disorder-specific treatments. The investigators propose Identity-Based Transdiagnostic Therapy (IBTT), a new treatment modality, to address the challenge of improving the outcomes of psychotherapy for young adults with anxiety and/or depression. IBTT is a psychological treatment for emotional disorders specifically designed for the youths in terms of their attitudes to treatment (attractiveness, engagement), by enhancing current constructivist psychotherapy practice with Explore Your Meanings (EYME), a technological platform including Virtual Reality (VR), to enable the immersive exploration of the participants self-identity. This project will allow testing the hypothesis that a novel brief psychotherapeutic intervention, IBTT, will be more efficacious in the treatment of the anxiety and/or depression of young adults than the well-established CBT-based Unified Protocol.

General objectives

With this project, the goal is to increase the efficacy of psychological therapies for anxiety and/or depression in young adults. That is, aiming to obtain better clinical results with IBTT, a promissory and novel treatment modality, than with the Unified Protocol, which is based on CBT and considered the most efficacious transdiagnostic treatment for emotional disorders. By obtaining supporting evidence for IBTT, the range of psychotherapeutic alternatives for these emotional disorders will be increased. This will benefit the potential for adapting the interventions to each patient's personal style, characteristics, and preferences. An optimal personalization of the treatment favors the patient's engagement in therapy and strengthens the therapeutic alliance, which, in turn, should be reflected in the facilitation of the change process.

Specific objectives

1. To assess the efficacy of an innovative VR-enhanced treatment modality of psychotherapy (IBTT) which has never been tested before. Differential outcomes will be considered not only in terms of statistical but also clinical significance, drop-out, and remission rates. In addition to the reduction of anxiety and depressive symptoms, our study is aimed at bettering psychological functioning, self-concept clarity, self-esteem, metacognitive mastery, well-being, and satisfaction with the services provided.
2. To identify baseline variables predicting outcome, including sociodemographic and clinical variables as well as characteristics of the personal construct system such as the level of cognitive conflict.
3. To gauge the significance of the therapeutic alliance in the two treatment modalities of the study, and its influence on the therapeutic outcomes.
4. To explore the personal views of participants concerning the therapy process that they will have experienced, as a way to advance our knowledge of the therapy process (including the incorporation of VR into that process) and of the potential adverse effects of each treatment. To compare this knowledge with the quantitative results of the study might be helpful for a better understanding of the entire process.
5. To analyze the gender-specific effects of the two treatments so that we can better adapt future applications of these treatments according to gender variables.
6. To disseminate the results of the project: the study protocol, therapy outcomes, the IBTT therapy manual, and the qualitative aspects.

Procedure

The project will be presented to clinical professionals of the centers participating in the study to stimulate the recruitment of participants according to the eligibility criteria. Referring professionals will provide a link (or QR) to participants interested in the study. Participants will find a welcome message with an explanation of the purpose and characteristics of the study and the option to provide informed consent to participate (including permission for the audio recording of the sessions). For those people who agree to participate, the online platform will ask to complete the sociodemographic data form, DASS-21, CORE-SFB, SCCS, RSES, MSAS-D, and LSS). After completion, an online meeting using a secure platform (Microsoft Teams) will be arranged for a clinical interview based on ICD-11 for diagnostic evaluation conducted by psychology graduates contracted by the project and trained for that purpose by researchers of the team. Participants meeting the inclusion criteria and not meeting any of the exclusion criteria will be randomly assigned to one of the two treatments of the study (1:1 ratio). Once the participant has completed the treatment (maximum 16 sessions), the end-of-therapy assessment will be conducted using DASS-21, CORE-SFB, SCCS, RSES, MSAS-D, and LSS. Then, a new online meeting will be arranged to administer the diagnostic interview and the Change Interview. It will be performed by the same evaluators who carried out the baseline assessment (whenever possible). A follow-up assessment including DASS-21, CORE-SFB, LSS, and CRES-4 will be conducted online three months after treatment termination.

Data analyses

Intention-to-treat analysis will be performed for the main statistical analyses. Descriptive analysis and intergroup comparisons will be performed with the Student´s T-test for quantitative variables, or the U-Mann-Whitney test for non-normally distributed data, and the Chi-square test for categorical variables. Linear mixed models will be used to analyze and compare treatment effects for the two arms. Baseline measurements, gender (coded as woman/male/other condition), and other sociodemographic and clinical variables will be entered into the model as covariates (DASS-21 as the primary outcome measure). For all the analyses, effect sizes and confidence intervals will be calculated.

Participants with comorbid conditions (eating and/or personality disorders, etc.) or taking psychotropic medication will not be excluded but they will be assessed and recorded for statistical analysis.

In addition to the statistical significance, the proportion of participants who attain clinically significant improvement on the outcome measures will be calculated and compared between treatment conditions. Clinical improvement will be calculated considering two conditions: reliable change (reliability of pre-to-post-difference score) and clinically significant change (to verify whether post-treatment scores lie in the normal or clinical range). To test the differences in frequencies between the treatment conditions, a Chi-square test will be applied.

The inclusion of CORE-SFB will permit assessment of the degree of therapeutic change with regard to psychological distress, psychosocial functioning, symptoms, and suicide risk. In addition, this application of CORE-SFB in each session will allow assessing the change experienced as a function of the number of sessions and the percentage of change session by session. Subgroup analyses by gender and other social determinants of health will be explored to check if there are significant differences in the therapy course. A secondary analysis will be performed by taking as a criterion variable satisfaction with life (LSS), as a way to assess the evolution of a positive outcome, and its relationship with the other outcomes will also be examined using correlational analysis. Other secondary analyses will examine the change that occurred in SCCS, RSES, and MSAS-D.

For the analysis of the Change Interview (used to capture the participants' subjective experience on the changes they may have experienced), the transcript of the audio recording of the interview will be used. Two independent researchers (psychology graduates) will record the mean number of changes elicited by subjects to be compared across samples, as well as the means of the following quantitative measures for each change, which are rated by respondents using a 5-point Likert scale: (1) relevance of the change experienced; (2) the extent to which the change was expected or surprising; (3) the extent to which the change was attributable to the effect of therapy. In addition, some qualitative analyses of the retrieved information will be conducted. First, two judges (psychology graduates) will independently perform content analysis, categorizing each change using the coding manual developed for this purpose. Second, another two judges (psychology graduates contracted) will also perform a similar analysis, but this time there will be no given categories, so these judges will have to make up their own. This second approach is based on the "grounded theory". This way, more information will be obtained about the areas of the subject's life that have been more affected by the occurring changes, as well as indicators of the techniques that were perceived as more useful.

ELIGIBILITY:
Inclusion Criteria:

• Participants with symptoms of depression and/or anxiety as their primary complaint.

Exclusion Criteria:

* Participants with post-traumatic stress, bipolar and substance use disorders, psychotic symptoms, organic brain dysfunction, marked suicidal ideation and/or intellectual disability.
* Participants receiving psychological treatment, unless it is suspended at the time of inclusion in the study itself in agreement with their therapist.
* Participants for whom the use of virtual reality may pose a risk, even a minor risk (epilepsia, acute otorhinolaryngological processes or recent interventions, severe cardiovascular disease, unstable hypertension, and pregnancy).
* Participants with substantial visual, hearing, and cognitive deficits.
* Participants who do not have enough competence to communicate in Spanish or Catalan.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scales (DASS-21) | DASS-21 will be administered at baseline, at 16 weeks (at completion), and at three-month follow-up.
  This 21-item version of the DASS comprises 7 items for its three scales (depression, anxiety, and stress) which are moderately correlated with each other. Respondents are asked to rate each item on a four-point Likert scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time) considering the past week.The scores for each scale range from 0 to 21 and the total score of the DASS-21 (0-63) is the primary outcome measure of the study. Higher scores in each scale indicate higher levels of depression, anxiety and stress, respectively.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation-Short Form B (CORE-SFB) | CORE-SFB will be administered at baseline, every session, at 16 weeks (at completion), and at three-month follow-up.
  CORE-SFB comprises 18 items (a short version of the 34-item self-report questionnaire CORE-OM) distributed across four scales assessing subjective well-being, symptoms or problems, life functioning, and risk. Respondents are asked to consider the past week and rate each item on a five-point Likert scale ranging from 0 (not at all) to 4 (most or all the time). Scores range between 0 and 72. Higher scores indicate worse outcome.
Session Rating Scale 3.0 (SRS 3.0) | Session Rating Scale 3.0 will be administered at the end of each therapy session, during 16 weeks.
  Session Rating Scale is a brief questionnaire designed to assess therapeutic alliance at the end of the session. It is composed of 4 items that have to be answered through a Visual Analog Scale (VAS) of 10 centimetres, and scores range between 0-40. Higher scores indicate greater appreciation of the relationship with the therapist, agreement with the therapist about the goals and issues discussed in the session, agreement with the therapist's method or approach, and global assessment of the session.
Life Satisfaction Scale (LSS) | Life Satisfaction Scale be administered at baseline, at 16 weeks (at completion), and at three-month follow-up.
  Life Satisfaction Scale is a single-item scale using a Likert scale of 10 points to capture the respondent's overall degree of satisfaction with life at the present moment. Scale ranging between 1 and 10. Higher scores indicate greater satisfaction.
Self-Concept Clarity Scale (SCCS) | SCCS will be administered at baseline and at 16 weeks (at completion).
  This version of the Self-Concept Clarity Scale consists of 12 items for assessing the level of clarity of the self-concept using a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores ranging between 12 and 60. Higher scores indicate stronger self-concept clarity.
Rosenberg Self-Esteem Scale (RSES) | Rosenberg Self-Esteem Scale will be administered at baseline and at 16 weeks (at completion).
  Rosenberg Self-Esteem Scale is a self-report instrument to measure global self-esteem and consists of 10 items using a four-item Likert scale ranging from 1 (strongly agree) to 4 (strongly disagree). Scores ranging between 10 and 40. Higher scores indicate greater self-judgment of value, confidence, and competence.
Metacognition Self-Assessment Scale, Subscale D (MSAS-5) | Metacognition Self-Assessment Scale (subscale D) will be administered at baseline and at 16 weeks (at completion).
  Metacognition Self-Assessment Scale (MSAS) is an 18-item self-report measure, answered on a five-point Likert scale (1 = never, 5 = always), range of 18-90 points, where higher scores indicate higher metacognitive performance. In this study, only the 5 items of the scale D of the MSAS. Scale D scores range of 5-25 points. Higher scores indicate greater metacognitive mastery, related to self-regulation and control activities.
Problem definition form | This form will be administered at baseline.
  This is a brief-structured interview aimed to define the problem (or the problems) the person is experiencing, its relevance, and the levels of distress it causes.
Change Interview | This form will be administered at 16 week (at completion)
  This semi-structured interview was created to assess the changes produced throughout therapy, the useful aspects, and the adverse effects of interventions from the patient's perspective.
Consumer Reports Effectiveness Scale (CRES-4) | Consumer Reports Effectiveness Scale only will be administered at three-month follow-up.
  To interpret Consumer Reports Effectiveness Scale-4, a score is considered that is on a scale ranging from 0 to 5 points. The higher the total score, the greater the satisfaction with the treatment according to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, PhD, Principal Investigator — University of Barcelona
Locations (2):
- Spain (2):
  - Badalona Serveis Assistencials, Badalona
  - Associació Centre Higiene Mental Nou Barris, Barcelona

REFERENCES:
- [Background] Barkham, M., Shapiro, D. A., & Morrison, L. (1988). Classification of psychological problems elicited by the Personal Questionnaire technique: A coding manual. Sheffield, UK: University of Sheffield, MRC/ESRC Social and Applied Psychology Unit.
- [Background] Campbell, J. D., Trapnell, P. D., Heine, S. J., Katz, I. M., Lavellee, L. F., y Lehman, D. R. (1996). Self-concept clarity: Measurement, personality correlates, and cultural boundaries. Journal of Personality and Social Psychology, 70, 141-156
- [Background] Carlucci L, Saggino A, Balsamo M. On the efficacy of the unified protocol for transdiagnostic treatment of emotional disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Jul;87:101999. doi: 10.1016/j.cpr.2021.101999. Epub 2021 Mar 9. PMID 34098412
- [Background] Duncan, B. L., Miller, S. D., Reynolds, L., Sparks, J., Claud, D., Brown, J. & Johnson, L. D. (2003). The session rating scale: Preliminary psychometric properties of a "working" alliance scale. Journal of Brief Therapy, 3(1), 3-12.
- [Background] Elliott, R., Slatick, E. & Urman, M. (2001). Qualitative change process research on psychotherapy: Alternative strategies. A: J. Frommer & D. L. Rennie (Eds.), Qualitative psychotherapy research: Methods and methodology (pp. 69-111). Pabst Science Publishers
- [Background] Elliott R, Wagner J, Sales CMD, Rodgers B, Alves P, Cafe MJ. Psychometrics of the Personal Questionnaire: A client-generated outcome measure. Psychol Assess. 2016 Mar;28(3):263-278. doi: 10.1037/pas0000174. Epub 2015 Jun 15. PMID 26075406
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Feixas, G., Pucurull, O., Roca, C., Paz, C., García-Grau, E., & Bados, A. (2012). Escala de Satisfacción con el tratamiento recibido (CRES-4): La versión en español. Revista de Psicoterapia, 89(23), 51-58.
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Lucas RE, Donnellan MB. Estimating the Reliability of Single-Item Life Satisfaction Measures: Results from Four National Panel Studies. Soc Indic Res. 2012 Feb 1;105(3):323-331. doi: 10.1007/s11205-011-9783-z. Epub 2011 Jan 13. PMID 23087538
- [Background] Marchette LK, Weisz JR. Practitioner Review: Empirical evolution of youth psychotherapy toward transdiagnostic approaches. J Child Psychol Psychiatry. 2017 Sep;58(9):970-984. doi: 10.1111/jcpp.12747. Epub 2017 May 26. PMID 28548291
- [Background] Pedone, R., Semerari, A., Riccardi, I., Procacci, M., Nicolò, G., & Carcione, A. (2017). Development of a self-report measure of metacognition: The metacognition self-assessment scale (MSAS). Instrument description and factor structure. Clinical Neuropsychiatry, 14(3), 185-194.
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton University Press